CLINICAL TRIAL: NCT04025918
Title: Closed-loop Double-vasopressor Automated System vs Manual Bolus Vasopressor to Treat Hypotension During Spinal Anaesthesia for Caesarean Section
Brief Title: Closed-loop Double-vasopressor Automated System to Treat Hypotension During Spinal Anaesthesia for Caesarean Section
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: KK Women's and Children's Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010/365/D
Record Dates: First submitted 2019-07-17; First posted 2019-07-19 (Actual); Last update posted 2019-07-19 (Actual); Status verified 2019-07

CONDITIONS: Hypotension
Keywords: hypotension; spinal anesthesia; cesarean section; phenylephrine; ephedrine; closed-loop system; continuous non-invasive monitor
MeSH Terms: conditions — Hypotension | interventions — Phenylephrine; Ephedrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vasopressor delivery automated system (Experimental): vasopressor delivery automated system that administered phenylephrine and ephedrine based on data from continuous non-invasive hemodynamic monitor
  Interventions: Device: Vasopressor automated delivery system; Drug: Phenylephrine; Drug: Ephedrine
- manual vasopressor delivery (Active Comparator): manual bolus that delivered phenylephrine and ephedrine based on data from non-invasive intermitted blood pressure monitor
  Interventions: Drug: Phenylephrine; Drug: Ephedrine; Device: Manual vasopressor delivery system

INTERVENTIONS:
Device: Vasopressor automated delivery system — Novel closed-loop system incorporating:
  1. Continuous non-invasive arterial pressure (CNAP) monitor that measured and recorded hemodynamic data in real time.
  2. Controller algorithm loaded onto a laptop computer that monitored the hemodynamic data from CNAP and determined if vasopressors should be administered.
  3. Two syringe pumps loaded with phenylephrine and ephedrine that was activated by the controller algorithm.
  Other Names: CNAP
  Arms: vasopressor delivery automated system
Drug: Phenylephrine — Phenylephrine is a vasopressor drug that was administered when the participant's systolic blood pressure fell below 90% of baseline systolic blood pressure, with heart rate of at least 60bpm.
Drug: Ephedrine — Ephedrine is a vasopressor drug that was administered when the participant's systolic blood pressure fell below 90% of baseline systolic blood pressure, with heart rate of less than 60bpm.
Device: Manual vasopressor delivery system — Manual dosing system consisting:
  1. Non-invasive intermittent blood pressure monitor that measured and recorded blood pressure at 1-minute intervals.
  2. Attending anesthesiologist that noted the blood pressure readings and manually administered phenylephrine or ephedrine according to the algorithm.
  Arms: manual vasopressor delivery

SUMMARY:
Hypotension occurs commonly during spinal anesthesia for caesarean section with maternal and fetal adverse effects. The investigators developed a double-vasopressor automated system incorporating continuous non-invasive arterial pressure monitoring (CNAP, CNSystems, Austria).

DETAILED DESCRIPTION:
Hypotension occurs commonly during spinal anesthesia for cesarean section with maternal and fetal adverse effects. The investigators developed a double-vasopressor automated system incorporating continuous non-invasive arterial pressure (CNAP, CNSystems, Austria) monitoring feeding hemodynamic data to a laptop computer, which triggers syringe pumps to deliver phenylephrine 50mcg or ephedrine 4mg (if heart rate<60 beats.min-1) every 30 seconds when systolic blood pressure fell to below 90% of baseline.

A randomised controlled trial was done to compare with manual bolus technique. With the manual bolus technique, phenylephrine 100mcg or ephedrine 8mg (if heart rate<60 beats.min-1) was given every 60 seconds by the attending anesthesiologist when systolic blood pressure was below 90% of baseline as measured by conventional intermittent non-invasive blood pressure monitoring.

ELIGIBILITY:
Inclusion Criteria:

* age 21-45 years old,
* weight 40-90 kg,
* height 145-170 cm

Exclusion Criteria:

* contraindications to spinal anaesthesia,
* allergy to drugs used in the study, and
* those with uncontrolled medical conditions such as hypertension, diabetes mellitus, and cardiovascular disease

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Study participants need to be pregnant and undergoing elective cesarean section
Enrollment: 216 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Hypotension | 1 day
  Incidence of systolic blood pressure less than 80% of baseline systolic blood pressure

SECONDARY OUTCOMES:
Hypertension | 1 day
  Incidence of systolic blood pressure more than 120% of baseline systolic blood pressure
Nausea and vomiting | 1 day
  Incidence of nausea and vomiting during cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Ban Leong Sng, FANZCA, Principal Investigator — KK Women's and Children's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ngan Kee WD. Prevention of maternal hypotension after regional anaesthesia for caesarean section. Curr Opin Anaesthesiol. 2010 Jun;23(3):304-9. doi: 10.1097/ACO.0b013e328337ffc6. PMID 20173633
- [Background] Sia AT, Tan HS, Sng BL. Closed-loop double-vasopressor automated system to treat hypotension during spinal anaesthesia for caesarean section: a preliminary study. Anaesthesia. 2012 Dec;67(12):1348-55. doi: 10.1111/anae.12000. Epub 2012 Sep 28. PMID 23020653
- [Result] Sng BL, Tan HS, Sia AT. Closed-loop double-vasopressor automated system vs manual bolus vasopressor to treat hypotension during spinal anaesthesia for caesarean section: a randomised controlled trial. Anaesthesia. 2014 Jan;69(1):37-45. doi: 10.1111/anae.12460. Epub 2013 Nov 20. PMID 24256483